CLINICAL TRIAL: NCT00782600
Title: A Phase 1, Randomized, 4-Period, 4-Sequence Cross-Over Study Of The Pharmacokinetics Of 3 Durations Of Release Of A Controlled Release Formulation And A Single Dose Of An Immediate Release Oral Suspension Of CE-224,535 In Normal Healthy Volunteers
Brief Title: Study of Controlled Release Formulations of CE-224,535 Against the Immediate Release Formulation in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A6341011
Record Dates: First submitted 2008-10-27; First posted 2008-10-31 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Pharmacokinetics Immediate Release Oral Suspension Controlled Release Formulation
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 mg oral suspension (Experimental): once daily for one day
  Interventions: Drug: suspension IR
- 50 mg CR Type 1 (Experimental): once daily for one day
  Interventions: Drug: CR 1
- 50 mg CR Type 2 (Experimental): once daily for one day
  Interventions: Drug: CR 2
- 50 mg SR Type 3 (Experimental): once daily for one day
  Interventions: Drug: CR 3

INTERVENTIONS:
Drug: suspension IR — 50 mg IR suspension once daily for one day
  Arms: 50 mg oral suspension
Drug: CR 1 — 50 mg shorter release CR once daily for one day
  Arms: 50 mg CR Type 1
Drug: CR 2 — 50 mg medium release CR once daily for one day
  Arms: 50 mg CR Type 2
Drug: CR 3 — longer release SR formulation once daily for one day
  Arms: 50 mg SR Type 3

SUMMARY:
This study is to test the idea that a controlled release formulation of CE-224,535 may allow for less frequent dosing and exposure to lower levels of drug than an immediate release formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs). A BMI lower limit of 17.5 kg/m2 may be rounded up to 18.0 kg/m2; a BMI upper limit of 30.5 kg/m2 may be rounded down to 30.0 kg/m2 and will be acceptable for inclusion.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.
* Any conHistory of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Various standard descriptive pharmacokinetics endpoints including: Cmin, Cmax, Tmax, AUC. | 1 month

SECONDARY OUTCOMES:
Safety laboratory testing including: blood electrolytes and liver and kidney function-related chemistries, complete blood counts, urinalysis, and electrocardiogram | 1 month
Other safety parameters including: physical examination and vital signs. | 1 month
Adverse Event Reporting as reported by subject and through investigator query and categorized by MedRA terminology. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6341011&StudyName=Study%20of%20%20Controlled%20Release%20Formulations%20of%20CE-224%2C535%20Against%20the%20Immediate%20Release%20Formulation%20in%20Normal%20Volunteers